CLINICAL TRIAL: NCT04038151
Title: Intuitive Control of a Hybrid Prosthetic Leg During Ambulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Levi Hargrove, Director, Regenstein Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00209522; 2R01HD079428-05 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-30 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Amputation
Keywords: Transfemoral Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condition A: Hybrid Leg (Experimental): Subject will be trained on use of the experimental device, the Hybrid Leg.
  Interventions: Device: Hybrid Leg
- Condition B: Passive Leg (Other): Subject will use their currently prescribed home passive prosthesis
  Interventions: Device: Prescribed Passive Prosthesis

INTERVENTIONS:
Device: Hybrid Leg — The Hybrid Knee uses an actively variable transmission in combination of a passive spring/damper system. This allows the motor torque output to be adapted to the requirements of active dynamic tasks - changing the effective transmission ration from zero (fully passive) for level ground walking to a maximum value (fully active) for sit-to-stand transfers. This provides physiological knee torque and speed with a small motor and primary transmission system while also maximizing electrical efficiency, which minimized battery weight. The knee prototype weights 1.7kg. The Semi-active ankle can actively reposition during non-weight bearing phases of gait and uses a non back driveable transmission to maintain its set point during weight bearing activities.
  Arms: Condition A: Hybrid Leg
Device: Prescribed Passive Prosthesis — Participants will participate in training sessions of community skills and advanced ambulation training for their home, prescribed passive prosthesis.
  Arms: Condition B: Passive Leg

SUMMARY:
The objective of this research is to determine the clinical benefits of an innovative and lightweight powered leg controlled using our intent recognition framework in laboratory and community environments.

DETAILED DESCRIPTION:
The hypothesis of this study is that using the Hybrid Leg with seamless, automatic transitions will result in participants choosing to become more active and improve their community participation compared to when using their own passive prosthetic leg.

The Hybrid Leg is an an innovative and lightweight powered leg that has 2 operating modes: active and passive. When in active mode, the Hybrid Leg is capable of supplying 120 NM of knee torque and actively repositioning the ankle during non-weight bearing phases of gait. When in passive mode, the motor and transmission are decoupled from the knee, which then behaves like an Ottobock 3R95 passive prosthetic knee, and the non-backdriveable mechanism of the ankle allows it to behave as an energy return foot. Allowing the device to behave passively if the battery becomes depleted or the actuators become damaged is an important enabling safety factor that will allow us to complete our study.

Phase 1: We will enroll 20 subjects a clinical trial of the leg and control system who will be fit with the Hybrid Leg and receive in-lab therapy to learn how to ambulate with the device.

Phase 2: Subjects will be randomized into a clinical trial of the leg and control system with an AB-BA design; condition A - subjects own device; condition B - Hybrid Leg. Subjects will complete an extensive ambulation and community mobility training to learn optimal use of their own passive device or the Hybrid Leg. After training the subjects will complete a full biomechanical analysis for each device as they complete ambulation circuits that include standing, level-ground walking, walking on slopes and on stairs, sit-stand transitions and transitions between these activities.

Phase 3: After completing phase 2 subjects will complete 4-week trials using their assigned prosthesis (Condition A or B) at home and within their community. During the trials subjects will be monitored using mobile phone based sensors and socket mounted activity monitor to determine how often the user performs the ambulation activities.

ELIGIBILITY:
Inclusion Criteria:

* A unilateral or bilateral lower limb amputation
* K2/K3/K4 ambulator with a prosthesis
* English speaking

Exclusion Criteria:

* Significant new injury that would prevent use of a prosthesis: The ability to consistently wear a prosthesis and perform activities of daily living and specific performance tasks is necessary to evaluate the relative benefits of the interventions.
* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data. The ability to obtain relevant user feedback through questionnaires and informal discussion adds significant value to this study.

  * Significant other comorbidity: Any other medical issues or injuries that would preclude completion of the study, use of the prostheses, or that would otherwise prevent acquisition of useable data by researchers.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Average daily number of steps | 4 weeks - data collected during 4 week home trial of each device, analyzed upon completion of 4 week home trial
  This outcome will be assessed using an accelerometery data measured using a mobile phone during the entire 4-week home trial of each device (Hybrid Leg and prescribed home device), resulting in a pair of outcomes for each subject. Statistical analysis will be done , first using a paired t-test (which assumes no carry-over and no device sequence effects), followed by the analysis using a linear mixed model with device and sequence group as fixed effects, and subject as the random effect. We expect that sequence will not be a statistically significant predictor, but that average daily steps will be significantly different between devices, with subjects taking significantly more steps when using the Hybrid Leg.
Average daily number of times subject switches between activities | 4 weeks - data collected during 4 week home trial of each device, analyzed upon completion of 4 week home trial
  This outcome will be assessed using an accelerometery data measured using a mobile phone during the entire 4-week home trial of each device (Hybrid Leg and prescribed home device), resulting in a pair of outcomes for each subject. Statistical analysis will be done , first using a paired t-test (which assumes no carry-over and no device sequence effects), followed by the analysis using a linear mixed model with device and sequence group as fixed effects, and subject as the random effect. We expect that sequence will not be a statistically significant predictor, but that average transitions will be significantly different between devices, with subjects taking significantly more transitioning between activities more when using the Hybrid Leg.

SECONDARY OUTCOMES:
10 Meter Walk Test | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  The 10mWT is used to assess walking speed in meters/second (m/s) over a short distance.
GPS tracking analysis | End of each 4 week home trial
  Subject-specific map of movement within the community will be generated and investigated for individual changes in community mobility and cross-referenced with their survey results. These data could provide insight into how well patient-reported measures reflect actual community participation, although this possibility is acknowledged to be exploratory
Six-Minute Walk Test | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  The 6MWT is a sub-maximal exercise test used to assess walking endurance and aerobic capacity. Participants will walk around the perimeter of a set circuit for a total of six minutes.
Hill Assessment Index | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  The Hill Assessment Index (HAI) is a 12 level ordinal scale developed to address different characteristics of hill ascent and descent in preparation comparing different prosthetic knee units. The HAI assesses gait patterns on hills combined with assistive device usage reflecting the quality of independence.
Stair Assessment Index | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  The Stair Assessment Index is a 14 level ordinal scale that assesses the functional ability of transfemoral amputees for stair ascent and descent. It is being used as a physical measurement tool to document different gait styles on the stairs.
Berg Balance Scale | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  The Berg Balance Scale is a 14 item objective measure that assesses static balance and fall risk in adults.
Functional Gait Assessment | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  The FGA is used to assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. The tool is a modification of the 8-item Dynamic Gait Index, developed to improve reliability and reduce ceiling effect.
5 Times Sit to Stand | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method of quantify functional lower extremity strength and /or identify movement strategies a patient used to complete transitional movements.
4 -Square Step Test | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  Test of dynamic balance that clinically assesses the person's ability to step over objects forward, sideways, and backwards.
Amputee Mobility Predictor | Lab visit prior to start of home trial and lab visit upon completion of 4 week trial with each device
  This instrument measures the ambulatory potential of lower limb amputees with and without the use of a prosthesis. It assesses the mobility of people with lower limb amputation prior to prosthetic fitting and predicts function following prosthetic prescription.

OTHER OUTCOMES:
Prosthesis Evaluation Questionnaire | Completion of each 4 week home trial
  The PEQ is a self-report questionnaire containing 54 questions that provide functional outcome measures in prosthetics that are more tuned to prosthesis related changes in quality of life.
Falls-Efficacy Scale | Completion of each 4 week home trial
  16 item self administered questionnaire designed to assess fear of falling in mainly community dwelling older population.
Orthotics and Prosthetics User Survey | Completion of each 4 week home trial
  The OPUS is a self report questionnaire consisting of five modules. It can be used for prosthetic and orthotic programs for quality assessment, to maintain awareness of improvement in activities, to evaluate changes in patients functional status and quality of lie and to assess satisfaction with devices and services.
World Health Organization Quality of Life Bref | Completion of each 4 week home trial
  The WHOQOL-BREF comprises 26 items which measure the following domains: physical health, psychological health, social relationships, and environment.

CONTACTS AND LOCATIONS:
Overall Officials: Levi Hargrove, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 2 years of study completion
Access Criteria: Data requests will be reviewed by the NU IRB and requester may need to sign a data access agreement.
URL: http://irb.northwestern.edu